CLINICAL TRIAL: NCT00151853
Title: Phase IV Study on the Efficacy of PPSB-SD and VP-VI in Patients Using Oral Anticoagulant Therapy and Undergoing Acute Cardiac Surgery With a Cardiopulmonary Bypass
Brief Title: Study Use of PPSB-SD and VP-VI in Patients With Anticoagulant Therapy and Undergoing Acute CPB Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Prothya Biosolutions (Industry)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAF2001.01
Record Dates: First submitted 2005-09-08; First posted 2005-09-09 (Estimated); Last update posted 2023-12-07 (Actual); Status verified 2006-01

CONDITIONS: CPB; Oral Anticoagulant Therapy
Keywords: CPB; oral anticoagulant therapy; plasma; PCC

INTERVENTIONS:
Drug: PPSB-SD

SUMMARY:
The purpose of this study was to study the efficacy of PPSB-SD and VP-VI in patients, who received anticoagulant treatment and who had to undergo acute cardiac surgery with a cardiopulmonary bypass (CPB).

DETAILED DESCRIPTION:
The value of oral anticoagulants such as coumarin derivatives as a therapy and in the prophylaxis of thrombosis is universally acknowledged. These medicinal products are used in the prevention of cerebral infarction, in patients with atrial fibrillation and in the secondary prevention of myocardial infarction. In case of elected surgery, the effect of coumarin derivatives can be reversed by a termination of the coumarin treatment and the administration of vitamin K orally, i.m. or i.v., which will restore the production of the vitamin K dependent coagulation factors. For patients due to undergo acute surgery, it will be unfavourable to await endogenous production of vitamin K dependent coagulation factor production.After CPB surgery, the patients need to be in a controlled coagulated state. Two products suitable to rapidly increase the concentration of vitamin K dependent coagulation factors, are fresh frozen plasma (FFP) and prothrombin complex concentrates (PCC). These products contain factor II, VII, IX and X and help to restore normal levels of the clotting fraction.Administration of these products prior to CPB surgery will decrease the INR to a level that is acceptable for surgery. In the Academic Hospital Leuven the standard procedure in cases of acute and elected CPB surgery is administration of VP-VI, a FFP-product made by OCTAPHARMA. In this study the standard treatment of 2x 400 ml VP-VI was compared with a treatment of PPSB Solvent Detergent® (PPSB-SD) according to the prescription regimen of CAF-DCF. PPSB-SD is a PCC product made by Sanquin Plasma Products (the Netherlands) for CAF-DCF (Belgium). The regimen as prescribed by CAF-DCF enables to calculate the quantity of PPSB-SD to administer on the basis of the patient's weight, the initial INR and the target INR. The expected outcome of the study was that in patients receiving PPSB-SD the target INR will be reached more frequently and more rapidly compared to patients receiving VP-VI.

ELIGIBILITY:
Inclusion Criteria:

age at least 18 years and due to undergo (semi-) acute cardiac surgery with a relatively stable haemodynamic condition.

and body weight less than 100 kg and informed consent and patients well controlled with acenocoumarol, phenprocoumon or warfarin.

-

Exclusion Criteria:

patients with an overdose of acenocoumarol, phenprocoumon or warfarin (INR > 7.8) and due to undergo (semi-) acute cardiac surgery hepatic insufficiency renal insufficiency anaphylactic reaction after administration of a blood product in the past disseminated intravascular coagulation (DIC) active thrombosis/pulmonary embolism intracardial thrombus patients treated with platelet inhibitors, except for aspirin (acetylsalicylic acid), who will be treated with aprotinine pregnancy breast-feeding

-

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-03; Study Completion 2004-09

PRIMARY OUTCOMES:
The primary objective of this study was to determine the mean time, median time and difference in time needed to reach the target INR of ≤1.5 after the end of CPB.

SECONDARY OUTCOMES:
The secondary objective of this study was to compare the number of post-(cpb)operative bleedings or re-operations for bleedings as well as the difference in the need of blood transfusions between the two groups

CONTACTS AND LOCATIONS:
Overall Officials: P FW Strengers, MD, Study Director — Prothya Biosolutions
Locations (1):
- University Hospital Gasthuisberg, Leuven, Belgium